CLINICAL TRIAL: NCT02105844
Title: Swiss Atrial Fibrillation Cohort Study - SWISS AF
Brief Title: Swiss Atrial Fibrillation Cohort Study
Acronym: SWISS-AF
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Medical Image Analysis Center (MIAC) Basel (Unknown); Schiller AG Baar (Unknown); Clinical Trial Unit, University Hospital Basel, Switzerland (Other); Cardiovascular Research Institute (CRIB) Basel (Unknown); Cardiocentro Ticino (Other)
Responsible Party: Sponsor
Other Study IDs: SWISS-AF
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; dementia; cognitive dysfunction; stroke; Magnetic resonance imaging
MeSH Terms: conditions — Atrial Fibrillation; Dementia; Cognitive Dysfunction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples with DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atrial Fibrillation: Cohort Study on patients with atrial fibrillation in Switzerland

SUMMARY:
Swiss-AF is a prospective observational, multicentric cohort study in Switzerland. Overall, 2600 patients with documented atrial fibrillation aged >65 years will be included and followed on a yearly basis.

Yearly clinical examinations include a detailed questionnaire on personal characteristics, a resting electrocardiogram, neurocognitive function tests and questionnaires on disability and quality of life. Blood sampling and brain magnetic resonance imaging are scheduled at baseline and after 2 years of follow-up.

The main study aims of this long term prospective study are to increase our knowledge on structural brain damage and its changes over time in patients with atrial fibrillation, to gain additional insights on the incidence and underlying mechanisms of cognitive decline in patients with atrial fibrillation and to evaluate the interrelationships of structural and functional brain damage in this population.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation documented within the last 24 months
* age >=45 years

Exclusion Criteria:

* acute illness
* inability to provide informed consent
* Only short episodes of reversible forms of atrial fibrillation

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 2415 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Stroke or systemic embolism | 2018 (after an average of 2.5 years of follow-up)

SECONDARY OUTCOMES:
Hospitalization for heart failure | 2018 (after an average of 2.5 years of follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Osswald, MD, Prof., Study Director — University Hospital, Basel, Switzerland; Michael Kuehne, MD, PD, exec. MBA, Principal Investigator — University Hospital, Basel, Switzerland; David Conen, MD MPH, Principal Investigator — McMaster University, Population Health Research Institute, Hamilton, Canada
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Kupper BC, Reiner MF, Werlen L, Aeschbacher S, Lee P, Allemann MS, Moschovitis G, Luscher T, Camici GG, Rodondi N, Adam L, Meyre PB, Bonati LH, Sinnecker T, Kuhne M, Osswald S, Conen D, Beer JH; Swiss-AF Investigators. Plasma beta-Thromboglobulin Is Inversely Associated With Cerebral Microbleeds in Atrial Fibrillation. Stroke. 2025 Dec;56(12):3414-3423. doi: 10.1161/STROKEAHA.124.049972. Epub 2025 Sep 17. PMID 40959897
- [Derived] Iten V, Herber E, Coslovsky M, Hennings E, Paladini RE, Reichlin T, Rodondi N, Muller AS, Stauber A, Beer JH, Brenner R, Conte G, Kobza R, Di Valentino M, Bedoya PC, Moradi F, Sinnecker T, Bonati LH, Kuhne M, Osswald S, Conen D, Aeschbacher S, Zuern CS; Swiss-AF and Beat-AF Investigators. Coffee consumption and adverse cardiovascular events in patients with atrial fibrillation. BMC Med. 2024 Dec 18;22(1):593. doi: 10.1186/s12916-024-03817-x. PMID 39696255
- [Derived] Barbagallo M, Springer A, Vanetta C, Allemann M, Lee P, Saeedi S, Aeschbacher S, Luciani M, Bonati LH, Moschovitis G, Scheu V, Rutishauser J, Kobza R, Di Valentino M, Meyre PB, Rodondi N, Conen D, Kuhne M, Osswald S, Beer JH; Swiss-AF investigators. Coffee Consumption Correlates With Better Cognitive Performance in Patients With a High Incidence for Stroke. J Am Heart Assoc. 2025 Jan 7;14(1):e034365. doi: 10.1161/JAHA.124.034365. Epub 2024 Dec 14. PMID 39673298
- [Derived] Carmine D, Aeschbacher S, Coslovsky M, Hennings E, Paladini RE, Peter R, Burger M, Reichlin T, Rodondi N, Muller AS, Ammann P, Conte G, Auricchio A, Moschovitis G, Bardoczi JB, Stauber A, De Perna ML, Zuern CS, Sinnecker T, Badertscher P, Sticherling C, Bonati LH, Conen D, Krisai P, Osswald S, Kuhne M. Blood pressure, brain lesions and cognitive decline in patients with atrial fibrillation. Front Cardiovasc Med. 2024 Sep 3;11:1449506. doi: 10.3389/fcvm.2024.1449506. eCollection 2024. PMID 39314770
- [Derived] Reiner MF, Bertschi DA, Werlen L, Wiencierz A, Aeschbacher S, Lee P, Rodondi N, Moutzouri E, Bonati L, Reichlin T, Moschovitis G, Rutishauser J, Kuhne M, Osswald S, Conen D, Beer JH. Omega-3 Fatty Acids and Markers of Thrombosis in Patients with Atrial Fibrillation. Nutrients. 2024 Jan 5;16(2):178. doi: 10.3390/nu16020178. PMID 38257071
- [Derived] Stauber A, Muller A, Rommers N, Aeschbacher S, Rodondi N, Bonati LH, Beer JH, Jeger RV, Kurz DJ, Liedtke C, Ammann P, Di Valentino M, Chocano P, Kobza R, Kuhne M, Conen D, Osswald S, Bernheim AM. Association of chocolate consumption with neurological and cardiovascular outcomes in atrial fibrillation: data from two Swiss atrial fibrillation cohort studies (Swiss-AF and BEAT-AF). Swiss Med Wkly. 2023 Aug 23;153:40109. doi: 10.57187/smw.2023.40109. PMID 37609948
- [Derived] Hennings E, Blum S, Aeschbacher S, Coslovsky M, Knecht S, Eken C, Lischer M, Paladini RE, Krisai P, Reichlin T, Rodondi N, Beer JH, Ammann P, Conte G, De Perna ML, Kobza R, Blum MR, Bossard M, Kastner P, Ziegler A, Muller C, Bonati LH, Pfister O, Zuern CS, Conen D, Kuhne M, Osswald S; Swiss-AF Investigators. Bone Morphogenetic Protein 10-A Novel Biomarker to Predict Adverse Outcomes in Patients With Atrial Fibrillation. J Am Heart Assoc. 2023 Mar 21;12(6):e028255. doi: 10.1161/JAHA.122.028255. Epub 2023 Mar 16. PMID 36926939
- [Derived] Luciani M, Muller D, Vanetta C, Diteepeng T, von Eckardstein A, Aeschbacher S, Rodondi N, Moschovitis G, Reichlin T, Sinnecker T, Wuerfel J, Bonati LH, Saeedi Saravi SS, Chocano-Bedoya P, Coslovsky M, Camici GG, Luscher TF, Kuehne M, Osswald S, Conen D, Beer JH; SWISS-AF Investigators. Trimethylamine-N-oxide is associated with cardiovascular mortality and vascular brain lesions in patients with atrial fibrillation. Heart. 2023 Feb 14;109(5):396-404. doi: 10.1136/heartjnl-2022-321300. PMID 36593094
- [Derived] Zwimpfer L, Aeschbacher S, Krisai P, Coslovsky M, Springer A, Paladini RE, Girod M, Hufschmid J, Knecht S, Badertscher P, Beer JH, Bonati LH, Zuern CS, Roten L, Reichlin T, Sticherling C, Conen D, Osswald S, Kuhne M. Neurocognitive function in patients with atrial fibrillation undergoing pulmonary vein isolation. Front Cardiovasc Med. 2022 Nov 25;9:1000799. doi: 10.3389/fcvm.2022.1000799. eCollection 2022. PMID 36505379
- [Derived] Girod M, Coslovsky M, Aeschbacher S, Sticherling C, Reichlin T, Roten L, Rodondi N, Ammann P, Auricchio A, Moschovitis G, Kobza R, Badertscher P, Knecht S, Krisai P, Marugg A, Aebersold H, Hennings E, Serra-Burriel M, Schwenkglenks M, Zuern CS, Bonati LH, Conen D, Osswald S, Kuhne M. Association of pulmonary vein isolation and major cardiovascular events in patients with atrial fibrillation. Clin Res Cardiol. 2022 Sep;111(9):1048-1056. doi: 10.1007/s00392-022-02015-0. Epub 2022 Apr 11. PMID 35403852
- [Derived] Rivolta MW, Mainardi LT, Laureanti R, Sassi R, Kuhne M, Rodondi N, Conte G, Moschovitis G, Schlageter V, Aeschbacher S, Conen D, Reichlin T, Roten L, Osswald S, Zuern CS, Auricchio A, Corino VDA. Association between ventricular repolarization parameters and cardiovascular death in patients of the SWISS-AF cohort. Int J Cardiol. 2022 Jun 1;356:53-59. doi: 10.1016/j.ijcard.2022.03.009. Epub 2022 Mar 9. PMID 35278571
- [Derived] Kuhne M, Krisai P, Coslovsky M, Rodondi N, Muller A, Beer JH, Ammann P, Auricchio A, Moschovitis G, Hayoz D, Kobza R, Shah D, Stephan FP, Schlapfer J, Di Valentino M, Aeschbacher S, Ehret G, Eken C, Monsch A, Roten L, Schwenkglenks M, Springer A, Sticherling C, Reichlin T, Zuern CS, Meyre PB, Blum S, Sinnecker T, Wurfel J, Bonati LH, Conen D, Osswald S; Swiss-AF Investigators. Silent brain infarcts impact on cognitive function in atrial fibrillation. Eur Heart J. 2022 Jun 6;43(22):2127-2135. doi: 10.1093/eurheartj/ehac020. PMID 35171989
- [Derived] Bano A, Rodondi N, Beer JH, Moschovitis G, Kobza R, Aeschbacher S, Baretella O, Muka T, Stettler C, Franco OH, Conte G, Sticherling C, Zuern CS, Conen D, Kuhne M, Osswald S, Roten L, Reichlin T; of the Swiss-Investigators. Association of Diabetes With Atrial Fibrillation Phenotype and Cardiac and Neurological Comorbidities: Insights From the Swiss-AF Study. J Am Heart Assoc. 2021 Nov 16;10(22):e021800. doi: 10.1161/JAHA.121.021800. Epub 2021 Nov 10. PMID 34753292
- [Derived] Hammerle P, Aeschbacher S, Springer A, Eken C, Coslovsky M, Dutilh G, Moschovitis G, Rodondi N, Chocano P, Conen D, Osswald S, Kuhne M, Zuern CS. Cardiac autonomic function and cognitive performance in patients with atrial fibrillation. Clin Res Cardiol. 2022 Jan;111(1):60-69. doi: 10.1007/s00392-021-01900-4. Epub 2021 Jun 22. PMID 34156525
- [Derived] Hammerle P, Eick C, Poli S, Blum S, Schlageter V, Bauer A, Rizas KD, Eken C, Coslovsky M, Aeschbacher S, Krisai P, Meyre P, Wuerfel J, Sinnecker T, Vesin JM, Beer JH, Moschovitis G, Bonati LH, Sticherling C, Conen D, Osswald S, Kuhne M, Zuern CS. Association of Heart Rate Variability With Silent Brain Infarcts in Patients With Atrial Fibrillation. Front Cardiovasc Med. 2021 May 21;8:684461. doi: 10.3389/fcvm.2021.684461. eCollection 2021. PMID 34095266
- [Derived] Benz AP, Aeschbacher S, Krisai P, Moschovitis G, Blum S, Meyre P, Blum MR, Rodondi N, Di Valentino M, Kobza R, De Perna ML, Bonati LH, Beer JH, Kuhne M, Osswald S, Conen D; BEAT-AF, Swiss-AF Investigators. Biomarkers of Inflammation and Risk of Hospitalization for Heart Failure in Patients With Atrial Fibrillation. J Am Heart Assoc. 2021 Apr 20;10(8):e019168. doi: 10.1161/JAHA.120.019168. Epub 2021 Apr 10. PMID 33843247
- [Derived] Reddiess P, Aeschbacher S, Meyre P, Coslovsky M, Kuhne M, Rodondi N, Baretella O, Beer JH, Kobza R, Moschovitis G, Di Valentino M, Muller C, Steiner F, Bonati LH, Sticherling C, Osswald S, Conen D; BEAT-AF and Swiss-AF investigators. Alcohol consumption and risk of cardiovascular outcomes and bleeding in patients with established atrial fibrillation. CMAJ. 2021 Jan 25;193(4):E117-E123. doi: 10.1503/cmaj.200778. PMID 33667180
- [Derived] Steiner F, Meyre PB, Aeschbacher S, Coslovsky M, Sinnecker T, Blum MR, Rodondi N, Cereda CW, di Valentino M, Wenger F, Cussigh A, Krisai P, Roten L, Reichlin T, Conen D, Osswald S, Bonati LH, Kuhne M; Swiss-AF Investigators. Association of the CHA2D(S2)-VASc Score and Its Components With Overt and Silent Ischemic Brain Lesions in Patients With Atrial Fibrillation. Front Neurol. 2021 Jan 12;11:609234. doi: 10.3389/fneur.2020.609234. eCollection 2020. PMID 33510705
- [Derived] Aeschbacher S, Blum S, Meyre PB, Coslovsky M, Vischer AS, Sinnecker T, Rodondi N, Beer JH, Moschovitis G, Moutzouri E, Hunkeler C, Burkard T, Eken C, Roten L, Zuern CS, Sticherling C, Wuerfel J, Bonati LH, Conen D, Osswald S, Kuhne M; Swiss-AF Investigators*. Blood Pressure and Brain Lesions in Patients With Atrial Fibrillation. Hypertension. 2021 Feb;77(2):662-671. doi: 10.1161/HYPERTENSIONAHA.120.16025. Epub 2020 Dec 28. PMID 33356398
- [Derived] Meyre PB, Springer A, Aeschbacher S, Blum S, Rodondi N, Beer JH, Di Valentino M, Ammann P, Blum M, Mathys R, Meyer-Zurn C, Bonati LH, Sticherling C, Schwenkglenks M, Kuhne M, Conen D, Osswald S; Swiss-AF investigators. Association of psychosocial factors with all-cause hospitalizations in patients with atrial fibrillation. Clin Cardiol. 2021 Jan;44(1):51-57. doi: 10.1002/clc.23503. Epub 2020 Nov 10. PMID 33169859
- [Derived] Hammerle P, Eick C, Blum S, Schlageter V, Bauer A, Rizas KD, Eken C, Coslovsky M, Aeschbacher S, Krisai P, Meyre P, Vesin JM, Rodondi N, Moutzouri E, Beer J, Moschovitis G, Kobza R, Di Valentino M, Corino VDA, Laureanti R, Mainardi L, Bonati LH, Sticherling C, Conen D, Osswald S, Kuhne M, Zuern CS; Swiss-AF Study Investigators. Heart Rate Variability Triangular Index as a Predictor of Cardiovascular Mortality in Patients With Atrial Fibrillation. J Am Heart Assoc. 2020 Aug 4;9(15):e016075. doi: 10.1161/JAHA.120.016075. Epub 2020 Jul 28. PMID 32750290
- [Derived] Gugganig R, Aeschbacher S, Leong DP, Meyre P, Blum S, Coslovsky M, Beer JH, Moschovitis G, Muller D, Anker D, Rodondi N, Stempfel S, Mueller C, Meyer-Zurn C, Kuhne M, Conen D, Osswald S; Swiss-AF Investigators. Frailty to predict unplanned hospitalization, stroke, bleeding, and death in atrial fibrillation. Eur Heart J Qual Care Clin Outcomes. 2021 Jan 25;7(1):42-51. doi: 10.1093/ehjqcco/qcaa002. PMID 31977016